CLINICAL TRIAL: NCT03278132
Title: A Phase IV Open-labelled, Single-centered, Stratified-randomized Clinical Trial in Zhejiang Province to Evaluate the Safety and Immunogenicity of EV71 Vaccine Developed by Sinovac Biotech Co., Ltd.
Brief Title: Phase IV Clinical Trial, Immunogenicity and Safety of EV71 Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Collaborators: Zhejiang Provincial Center for Disease Control and Prevention (Other Government); Shangyu District Center for Disease Control and Prevention (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-EV71-4011
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: Inactivated Enterovirus Type 71 (EV71) Vaccine; Safety; Immunogenicity; Infant
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EV71 vaccine & blood sampling (0, 10,60) (Experimental): This group receive two doses injection of EV71 vaccine (0, 28 days), and three times of blood sampling on day of 0, 10, and 60 respectively for EV71 neutralizing antibody detection.
  Interventions: Biological: EV71 vaccine
- EV71 vaccine & blood sampling (0, 20,60) (Experimental): This group receive two doses injection of EV71 vaccine (0, 28 days), and three times of blood sampling on day of 0, 20, and 60 respectively for EV71 neutralizing antibody detection.
  Interventions: Biological: EV71 vaccine
- EV71 vaccine& blood sampling (0, 30, 60) (Experimental): This group receive two doses injection of EV71 vaccine (0, 28 days), and three times of blood sampling on day of 0, 30, and 60 respectively for EV71 neutralizing antibody detection.
  Interventions: Biological: EV71 vaccine

INTERVENTIONS:
Biological: EV71 vaccine — Two doses vaccination of EV71vaccine (Intramuscular injection, 0.5ml) with a schedule of 0, 28 days.

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of EV71 vaccine in infants aged 6 to 35 months old, by detecting the dynamic changes of neutralizing antibody at different time after vaccination

DETAILED DESCRIPTION:
This study is an open-labelled, single-centered, stratified-randomized, phase IV clinical trial. The purpose of this study is to evaluate the immunogenicity and safety of EV71 vaccine (developed by Sinovac Biotech Co., Ltd.) in infants aged 6 to 35 months old, by detecting the dynamic changes of neutralizing antibody at different times after vaccination. The enrolled subjects in this study receive two doses of EV71 vaccine with 1-month interval between doses. To evaluate safety of the vaccine, subjects will be observed for 30 days after the injection for the potential adverse events. To evaluate the immunogenicity of the vaccine, venous blood will be collected for the neutralizing antibody detection prior to vaccination, 10/20/30 days after the 1st dose and 30 days after the 2nd dose vaccination. All subjects will receive blood sampling for three times. Subjects will be randomly assigned to receive blood sampling at 10/20/30 days after 1st dose injection, with a ratio of 1: 1: 1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 6-35 months old
* Guardian(s) of the volunteer should be capable of understanding the written consent form, and such form should be signed before the infant being included into this study
* Proven legal identity

Exclusion Criteria:

For subjects with any of the following conditions, vaccination should not be administrated:

* History of hand foot and mouth disease
* Allergy to gentamicin; history of allergy to any vaccine or vaccine ingredient, or serious adverse reaction(s) to vaccination, such as urticaria, difficulty in breathing, angioneurotic edema, pain, etc
* Severe chronic diseases
* Thrombocytopenia or hemorrhagic disease
* Immunodeficiency disease or receipt of immunosuppressant treatment
* Uncontrolled epilepsy or progressive neurological disorders(e.g. Guillain-Barre syndrome)
* Acute disease or acute stage of chronic disease prior to the study entry
* History of thyroidectomy, thyroid disease within 12 months prior to the study entry
* Asplenia or functional asplenia
* Axillary temperature >37.0 ℃
* Any other factor that suggesting the volunteer is unsuitable for this study based on the judgment of investigators

Exclusion Criteria of the Second Injection:

* Subjects with any of the following conditions are forbidden to continue the 2nd dose of vaccination:

  1. Any serious adverse event that has a causal relationship with the investigated vaccine
  2. Severe allergic reactions or hypersensitivity after vaccination (including urticaria / rash appear within 30 minutes after vaccination
  3. Any confirmed or suspected autoimmune disease or immunodeficiency disease (e.g., HIV infection)
  4. Other reactions (including severe pain, severe swelling, severe activity limitation, persistent hyperthermia, severe headache or other systemic or local reactions)determined by the investigators
* For subjects suffering from acute disease or acute stage of chronic disease , whether to continue vaccination depends on themselves
* Subjects with the following conditions may receive vaccination in delayed time or withdraw from the study depending on the judgment of investigator

  1. Acute disease (moderate or severe disease with or without fever) in case of vaccination
  2. Axillary temperature > 37.0 °C

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2017-07-16 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
The seroconversion rate of EV71 neutralizing antibody 30 days after the two doses vaccination | 30 days
  Immunogenicity indicator

SECONDARY OUTCOMES:
The seroconversion rate of EV71 neutralizing antibody 10, 20 and 30 days after the first dose vaccination | 10,20,and 30 days
  Immunogenicity indicator
The seropositive rate of EV71 neutralizing antibody 10, 20, 30, and 60 days after the first dose vaccination | 10, 20,30,and 60 days
  Immunogenicity indicator
GMT and GMT increase fold of EV71 neutralizing antibody 10,20,30,and 60 days after the first dose vaccination | 10,20，30，and 60 days
  Immunogenicity indicator
Incidence of unsolicited local or systemic adverse events within 3 days after each dose | 3 days
  Safety indicator
Incidence of unsolicited adverse events within 30 days after each dose | 30 days
  Safety indicator
Incidence of the serious adverse events within 60 days after the first dose vaccination | 60 days
  Safety indicator

CONTACTS AND LOCATIONS:
Overall Officials: Huakun Lv, Principal Investigator — Zhejiang Provincial Center for Disease Control and Prevention
Locations (1):
- Shangyu District Center for Disease Control and Prevention, Shaoxing, Zhejiang, China

REFERENCES:
- [Derived] Wang S, Zeng J, Zhang X, Gan Z, Fan J, Chen Y, Liang Z, Hu X, Zeng G, Lv H. Short-term dynamic changes in neutralizing antibodies against enterovirus 71 after vaccination. Hum Vaccin Immunother. 2020 Jul 2;16(7):1595-1601. doi: 10.1080/21645515.2020.1711678. Epub 2020 Jan 24. PMID 31977278